CLINICAL TRIAL: NCT00766532
Title: Do Aromatase Inhibitors (AIs) Decrease Intestinal Calcium Absorption?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2008-0144
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer; Osteoporosis; Osteopenia; Fracture
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis; Bone Diseases, Metabolic; Fractures, Bone | interventions — Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aromatase inhibitor therapy (Experimental): aromatase inhibitor therapy for six weeks
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Aromatase Inhibitor — Any aromatase inhibitor started as initial adjuvant therapy

SUMMARY:
Research Question: Do Aromatase Inhibitors Decrease Intestinal Calcium Absorption?

Study Design: Postmenopausal women with early stage breast cancer initiating aromatase inhibitor adjuvant therapy will participate in this two-month study. The primary study outcome is the change in intestinal calcium absorption following such therapy. Secondary outcomes are the changes in bone resorption markers and musculoskeletal signs and symptoms after initiation of therapy.

We will interview women and review their medical records to determine eligibility. Eligible subjects will undergo two calcium absorption studies. The first study will determine their baseline calcium absorption, and the second study will occur after taking an aromatase inhibitor daily for at least 6 weeks. Women will present to the research unit in the early morning and receive an oral and intravenous stable calcium tracer with breakfast. Over the next 24 hours, we will collect all urine for measurement of its calcium content. During each inpatient stay, we will assess musculoskeletal symptoms by questionnaire and joint examination. Each woman will complete a four-day diet diary twice during the study.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 5 years past menopause, defined as date of last menses or bilateral oophorectomy
* Newly diagnosed breast cancer and starting an AI as initial adjuvant therapy

Exclusion Criteria

* Recent, current or planned chemotherapy for breast cancer, as this may have independent effects on intestinal health, calcium homeostasis and bone turnover
* Allergy or intolerance to orange juice, as one isotope is given with orange juice
* Current use of over-the-counter or prescription antacids, as they may influence Ca-Ab
* Intestinal conditions associated with malabsorption or low gastric acid levels including Crohn's disease, ulcerative colitis, pernicious anemia, bacterial overgrowth, celiac sprue, chronic diarrhea or use of antibiotics within the past month
* Known Stage 4 or 5 Chronic Kidney Disease, defined as an estimated GFR <30 cc/minute
* Use of medications known to interfere with calcium or vitamin D metabolism, including oral steroids or anticonvulsants
* Significant lymphedema precluding adequate intravenous access

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Result] Tevaarwerk A, Burkard ME, Wisinski KB, Shafer MM, Davis LA, Gogineni J, Crone E, Hansen KE. Aromatase inhibitors and calcium absorption in early stage breast cancer. Breast Cancer Res Treat. 2012 Jul;134(1):245-51. doi: 10.1007/s10549-012-1982-z. Epub 2012 Feb 18. PMID 22350731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with early stage breast cancer and planning to start aromatase inhibitor therapy.
Pre-assignment Details: Participants completed a four-day food diary
Groups:
- Arm Title- Aromatase Inhibitor Therapy: calcium absorption was measured among subjects at baseline and after taking aromatase inhibitor therapy.
Period: Overall Study
Arm/Group | Arm Title- Aromatase Inhibitor Therapy
Started | 12
Completed | 10
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Intestinal Calcium Absorption Related to Aromatase Inhibitor Therapy
Description: intestinal calcium absorption
Time Frame: baseline and 6 weeks later
Population: 12 subjects provided informed consent but two dropped and did not undergo calcium absorption study visits. 10 subjects completed all calcium absorption study visits.
Measure: Mean (Standard Deviation); unit: percent calcium absorption
Arm/Group | Aromatase Inhibitor Therapy
Number analyzed (Participants) | 10
percent calcium absorption | 16 (6)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No